CLINICAL TRIAL: NCT01548274
Title: Impact of Sarpogrelate in the Function of Endothelial Progenitor Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aichi Gakuin University (Other)
Responsible Party: Principal Investigator, Keiko Naruse, Associate professor, Aichi Gakuin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGU-65
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Atherosclerosis
Keywords: endothelial progenitor cells
MeSH Terms: conditions — Atherosclerosis | interventions — sarpogrelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sarpogrelate — Sarpogrelate 300mg/day

SUMMARY:
The purpose of this study is to evaluate the effects of Sarpogrelate in endothelial progenitor cells of patients with atherosclerosis.

DETAILED DESCRIPTION:
Endothelial progenitor cells play an important role in vasculogenesis and vascular repair. Sarpogrelate, a inhibitor of HT2A, is used an an anti-platelet drug, however, a direct effect in vascular cells is supposed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerosis

Exclusion Criteria:

* Patients with high risk of bleeding
* Patients with pregnancy
* Patients with allergic reaction of Salpogrelate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The number and function of endothelial progenitor cells | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Aichi-Gakuin University, Nagoya, Aichi-ken, Japan